CLINICAL TRIAL: NCT05493761
Title: Effect of Anti-osteoporotic Medications on Hepatic Steatosis and Fibrosis of Women With Postmenopausal Osteoporosis and Nonalcoholic Fatty Liver Disease
Brief Title: Effect of Anti-osteoporotic Medications on Nonalcoholic Fatty Liver Disease
Acronym: OsteoNAFLD
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: 424 General Military Hospital (Other)
Responsible Party: Principal Investigator, Stergios A Polyzos, Associate Professor of Pharmacology, Aristotle University Of Thessaloniki
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 88235
Record Dates: First submitted 2022-07-24; First posted 2022-08-09 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Nonalcoholic Fatty Liver; Osteoporosis, Postmenopausal
Keywords: nonalcoholic fatty liver disease; hepatic steatosis; hepatic fibrosis; bisphosphonates; denosumab; postmenopausal osteoporosis; treatment; alendronate; nonalcoholic steatohepatitis; NAFLD; NASH; elastography; metabolic dysfunction-associated steatotic liver disease; metabolic dysfunction-associated steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Osteoporosis, Postmenopausal; Fatty Liver; Liver Cirrhosis | interventions — Denosumab; Alendronate

STUDY DESIGN:
Intervention Model Description: Multicenter, non-randomized, non-blinded, parallel group, one-year clinical trial
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- "Denosumab" (Experimental): 35 postmenopausal women with low bone mineral density (BMD) and NAFLD will receive denosumab.
  Interventions: Drug: Denosumab
- "Alendronate" (Active Comparator): 35 postmenopausal women with low bone mineral density (BMD) and NAFLD will receive alendronate.
  Interventions: Drug: Alendronate Sodium

INTERVENTIONS:
Drug: Denosumab — 60 mg (1ml) administered subcutaneously once every 6 months for 12 months (totally 2 injections). Patients will also be supplemented with calcium carbonate (1000 mg/d) and cholecalciferol (800 IU/day), according to the recent guidelines.
  Other Names: Prolia
  Arms: "Denosumab"
Drug: Alendronate Sodium — 70 mg (1 tablet) administered per os once weekly for 12 months. Patients will also be supplemented with calcium carbonate (1000 mg/d) and cholecalciferol (800 IU/day), according to the recent guidelines.
  Other Names: Fosamax
  Arms: "Alendronate"

SUMMARY:
Nonalcoholic fatty liver disease (NAFLD) is a chronic, metabolic liver disease that is closely related to obesity, type 2 diabetes mellitus (T2DM) and metabolic syndrome (MetS) in a bidirectional mode. NAFLD affects approximately 25% of the worldwide population. NAFLD refers to a phenotypic spectrum, including steatosis, inflammation and fibrosis, which can lead to cirrhosis and hepatocellular carcinoma in a minority of patients. However, despite its high prevalence, morbidity and mortality, as well as the extensive research in the field, there is not to-date a licensed medication specifically for NAFLD.

Emerging evidence supports a potential association between NAFLD and osteoporosis; the prevalence of osteoporosis is probably higher in patients with NAFLD and, vise versa, the prevalence of NAFLD may be higher in patients with osteoporosis. In this context, it has been proposed that certain medications for osteoporosis may also prove to be beneficial to NAFLD.

Denosumab, a human monoclonal IgG2 antibody against the receptor activator of nuclear factor kappa-B (NF-κB) ligand (RANKL), is currently an established treatment for osteoporosis and other metabolic bone diseases. The axis RANKL-receptor activator of nuclear factor NF-κB (RANK)-osteoprotegerin (OPG) has been demonstrated as a key regulator of bone metabolism and, when dysregulated, it contributes to the pathogenesis of osteoporosis and other metabolic bone diseases. Interestingly, experimental studies have shown that circulating and hepatic RANKL may be upregulated in mice with diet-induced NAFLD, rendering RANKL a potential contributor to the pathogenesis of NAFLD, and ideally, a promising pharmacological target.

On the other hand, bisphosphonates, another established, first-line treatment for osteoporosis, are expected to have no significant effect on hepatic metabolism in patients with NAFLD due to their pharmacokinetics and mechanism of action.

This is a prospective non-randomized study which aims to investigate the comparative effect of denosumab versus bisphosphonates on hepatic steatosis and fibrosis in women with postmenopausal osteoporosis and concomitant NAFLD.

ELIGIBILITY:
Inclusion Criteria:

* postmenopausal women aged > 40 years
* diagnosis of osteoporosis, or osteopenia and Fracture Assessment Risk (FRAX) score indicative for initiation of anti-osteoporotic treatment, or osteopenia and history of low-energy fracture. Evaluation of osteopenia and osteoporosis will be based on bone mineral density (BMD) of the lumbar spine and/or the femoral neck of the non-dominant hip measured with dual energy X-ray absorptiometry (DXA)
* diagnosis of NAFLD based on non-invasive indices of hepatic steatosis
* written informed consent

Exclusion Criteria:

* mean ethanol consumption >10 g/day
* a history of other chronic liver disease (e.g., viral hepatitis, autoimmune hepatitis, primary sclerosing cholangitis, primary biliary cholangitis and overlap syndromes, drug-induced liver injury, hemochromatosis, Wilson's disease, α1-antitrypsin deficiency)
* liver cirrhosis
* any malignancy
* chronic kidney disease
* uncontrolled hypothyroidism or hyperthyroidism
* use of the following medications within a 12-month period before baseline associated with drug-induced fatty liver: interferon, tamoxifen, amiodarone, aloperidin, glucocorticosteroids, anabolic steroids, any medication against tuberculosis, epilepsy or viruses, methotrexate, parenteral nutrition
* use of the following medications within a 12-month period before baseline associated probably with improvement in fatty liver: vitamin E, pioglitazone, insulin, glucagon-like peptide-1 receptor agonists (GLP-1RAs), sodium-glucose co-transporter-2 inhibitors (SGLT-2), orlistat, ursodeoxycholic acid
* use of any anti-osteoporotic medication within a 12-month period before baseline, except for calcium and vitamin D

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 72 (Actual)
Dates: Start 2022-12-23 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Hepatic steatosis: Ultrasound-Guided Attenuation Parameter (UGAP) measured on an ultrasound machine GE Logiq E10s. | 12 months
  1. Between-within group interactions in UGAP (baseline to endpoint)
  2. Between groups difference in change in UGAP (baseline to endpoint)
  UGAP is a non-invasive index based on the attenuation quantification of the ultrasound beam through the hepatic parenchyma, thus used for hepatic steatosis quantification. Cut-off values of > 0.53 dB/cm/MHz, >0.60 dB/cm/MHz, and >0.65 dB/cm/MHz have been proposed for the diagnosis of steatosis grade S1, S2, and S3, respectively.

SECONDARY OUTCOMES:
Hepatic fibrosis: liver stiffness (LS) measured with 2D Shear Wave Elastography (2D SWE) on an ultrasound machine GE Logiq E10s. | 12 months
  1. Between-within group interactions in LS (baseline to endpoint)
  2. Between groups difference in change in LS (baseline to endpoint)
  2D SWE is a non-invasive tool measuring the hepatic parenchyma stiffness, thus indirectly suggesting fibrosis stage (F). Cut-offs values of <8.27 kPa, 8.27-9.39 kPa, 9.40-11.88 kPa and >11.88 kPa have been proposed for F0-F1, F2, F3, and F4, respectively.
Hepatic steatosis non-invasive index: Fatty Liver Index (FLI). | 12 months
  1. Between-within group interactions in FLI (baseline to endpoint)
  2. Between groups difference in changes in FLI (baseline to endpoint)
  FLI is a non-invasive hepatic steatosis index, which is based on BMI, waist circumference, GGT and triglycerides. FLI ≥60 is associated with the presence of steatosis, while FLI <30 rules out the presence of steatosis.
Hepatic steatosis non-invasive index: Hepatic Steatosis Index (HSI). | 12 months
  1. Between-within group interactions in HSI (baseline to endpoint)
  2. Between groups difference in changes and HSI (baseline to endpoint)
  HSI is a non-invasive hepatic steatosis index, which is based on AST, ALT, BMI, gender and the presence or not of T2DM. HSI ≥36 is associated with the presence of steatosis, while HSI <30 rules out the presence of steatosis.
Hepatic fibrosis non-invasive index: NAFLD fibrosis score (NFS). | 12 months
  1. Between-within group interactions in NFS (baseline to endpoint)
  2. Between groups difference in changes in NFS (baseline to endpoint)
  NFS is a non-invasive hepatic fibrosis index, which is based on age, BMI, AST, ALT, platelets, albumin and the presence or not of T2DM. NFS >0.675 is associated with high probability of advanced hepatic fibrosis (F3-F4), while NFS <-1.455 is associated with low probability of advanced hepatic fibrosis (F3-F4).
Hepatic fibrosis non-invasive index: Fibrosis-4 index (FIB-4). | 12 months
  1. Between-within group interactions in FIB-4 (baseline to endpoint)
  2. Between groups difference in changes in FIB-4 (baseline to endpoint)
  FIB-4 is a non-invasive hepatic fibrosis index, which is based on age, AST, ALT and platelets. FIB-4 ≥2.67 is associated with high probability of advanced hepatic fibrosis (F3-F4), while FIB-4 <1.3 (when age <65 years) or <2.0 (when age ≥65 years) is associated with low probability of advanced hepatic fibrosis (F3-F4).
Hepatic fibrosis non-invasive index: AST-to-Platelet Ratio Index (APRI). | 12 months
  1. Between-within group interactions in APRI (baseline to endpoint)
  2. Between groups difference in changes in APRI (baseline to endpoint)
  APRI is a non-invasive hepatic fibrosis index, which is based on AST, ALT and platelets. APRI ≥1 is associated with high probability of advanced hepatic fibrosis (F3-F4), while APRI <0.5 is associated with low probability of advanced hepatic fibrosis (F3-F4).
Liver function tests: alanine aminotransferase (ALT). | 12 months
  Between-within group interactions in ALT (baseline to endpoint)
  The normal range for ALT is 4-36 U/L, but it may be different in different laboratories. Higher values may indicate hepatocellular injury.
Liver function tests: aspartate aminotransferase (AST) | 12 months
  Between-within group interactions in AST (baseline to endpoint)
  The normal range for AST is 8-33 U/L, but it may be different in different laboratories. Higher values may indicate hepatocellular injury.
Insulin resistance index: Homeostasis Model Assessment - Insulin Resistance (HOMA-IR) | 12 months
  Between-within group interactions in HOMA-IR (baseline to endpoint)
  HOMA-IR is calculated by the formula: fasting glucose (mg/dl) × insulin (mU/L)/405, and indicates the degree of insulin resistance; higher scores indicate greater insulin resistance. A HOMA-IR value ≥2.5 is indicative of insulin resistance.
Lipid profile: total cholesterol | 12 months
  Between-within group interactions in total cholesterol (baseline to endpoint)
  Total cholesterol levels <200mg/dl are considered acceptable, 200-239 mg/dl are borderline high, and ≥240 mg/dl are considered high; however, these cut-offs differentiate according to other cardiovascular risk factors.
Lipid profile: triglycerides | 12 months
  Between-within group interactions in triglycerides (baseline to endpoint)
  Triglycerides levels <150mg/dl are considered acceptable, 150-199 mg/dl are borderline high, and ≥200 mg/dl are considered high.
Lipid profile: low-density lipoprotein cholesterol (LDL-C) | 12 months
  Between-within group interactions in LDL-C (baseline to endpoint)
  LDL-C levels <100mg/dl are considered optimal, 100-129 mg/dl are borderline high, and >130 mg/dl are considered high; however, these cut-offs differentiate according to other cardiovascular risk factors.
Lipid profile: high-density lipoprotein cholesterol (HDL-C) | 12 months
  Between-within group interactions in HDL-C (baseline to endpoint)
  For women, the normal range for HDL-C is 50-90 mg/dl. Higher HDL-C are regarded as better.
Serum adipokines: leptin | 12 months
  Between-within group interactions in leptin (baseline to endpoint)
  For women, the normal range for leptin is 5-15 ng/ml, but it may be different for different ELISA kits.
Serum adipokines: adiponectin | 12 months
  Between-within group interactions in adiponectin (baseline to endpoint)
  The normal range for adiponectin is 5-30 μg/ml, but it may be different for different ELISA kits.

CONTACTS AND LOCATIONS:
Overall Officials: Ilias D Vachliotis, MD, PhDc, Study Director — School of Medicine, Aristotle University of Thessaloniki; Athanasios D Anastasilakis, MD, PhD, Study Director — 424 General Military Hospital, Thessaloniki, Greece; Antonis Goulas, MD, PhD, Study Director — School of Medicine, Aristotle University of Thessaloniki; Dimitrios G Goulis, MD, PhD, Study Director — School of Medicine, Aristotle University of Thessaloniki; Stergios A Polyzos, MD, PhD, Principal Investigator — School of Medicine, Aristotle University of Thessaloniki; Zoe A Efstathiadou, MD, PhD, Study Director — Department of Endocrinology, "Hippokration" General Hospital of Thessaloniki; Vasileios Rafailidis, MD, PhD, Study Director — School of Medicine, Aristotle University of Thessaloniki
Locations (3):
- Greece (3):
  - Department of Endocrinology, "Hippokration" General Hospital of Thessaloniki, Thessaloniki
  - 1st Department of Obstetrics and Gynecology, School, of Medicine, Aristotle University of Thessaloniki, Thessaloniki
  - 424 General Military Hospital, Thessaloniki

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make IPD and related data dictionaries available
Supporting Information: Study Protocol, SAP
Time Frame: 12 months after the publication of the study.
Access Criteria: Yet unknown

REFERENCES:
- [Background] Makri E, Goulas A, Polyzos SA. Epidemiology, Pathogenesis, Diagnosis and Emerging Treatment of Nonalcoholic Fatty Liver Disease. Arch Med Res. 2021 Jan;52(1):25-37. doi: 10.1016/j.arcmed.2020.11.010. Epub 2020 Dec 14. PMID 33334622
- [Background] Polyzos SA, Goulas A. Treatment of nonalcoholic fatty liver disease with an anti-osteoporotic medication: A hypothesis on drug repurposing. Med Hypotheses. 2021 Jan;146:110379. doi: 10.1016/j.mehy.2020.110379. Epub 2020 Nov 7. PMID 33208241
- [Background] Filip R, Radzki RP, Bienko M. Novel insights into the relationship between nonalcoholic fatty liver disease and osteoporosis. Clin Interv Aging. 2018 Oct 4;13:1879-1891. doi: 10.2147/CIA.S170533. eCollection 2018. PMID 30323574
- [Background] Anastasilakis AD, Polyzos SA, Makras P. THERAPY OF ENDOCRINE DISEASE: Denosumab vs bisphosphonates for the treatment of postmenopausal osteoporosis. Eur J Endocrinol. 2018 Jul;179(1):R31-R45. doi: 10.1530/EJE-18-0056. Epub 2018 Apr 24. PMID 29691303
- [Background] Zhong L, Yuan J, Huang L, Li S, Deng L. RANKL Is Involved in Runx2-Triggered Hepatic Infiltration of Macrophages in Mice with NAFLD Induced by a High-Fat Diet. Biomed Res Int. 2020 May 25;2020:6953421. doi: 10.1155/2020/6953421. eCollection 2020. PMID 32596356
- [Background] Rinotas V, Niti A, Dacquin R, Bonnet N, Stolina M, Han CY, Kostenuik P, Jurdic P, Ferrari S, Douni E. Novel genetic models of osteoporosis by overexpression of human RANKL in transgenic mice. J Bone Miner Res. 2014;29(5):1158-69. doi: 10.1002/jbmr.2112. PMID 24127173
- [Background] Vachliotis ID, Anastasilakis AD, Goulas A, Goulis DG, Polyzos SA. Nonalcoholic fatty liver disease and osteoporosis: A potential association with therapeutic implications. Diabetes Obes Metab. 2022 Sep;24(9):1702-1720. doi: 10.1111/dom.14774. Epub 2022 Jun 14. PMID 35589613